CLINICAL TRIAL: NCT07214454
Title: An Open Label, Single-site Feasibility Study of Transcranial Direct Current Stimulation (tCDS), Using the Nettle Device, for the Treatment of Chronic Migraine.
Brief Title: TCDS for the Treatment of Chronic Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 361355
Record Dates: First submitted 2025-09-30; First posted 2025-10-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Migraine Headache; Transcranial Direct Current Stimulation
Keywords: chronic migraine treatment; transcranial direct current stimulation; non-invasive neuromodulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Open label, single site, feasibility study of transcranial direct current stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with transcranial direct current stimulation (Experimental): Patients will complete three months treatment of 20 minutes daily use of the Nettle device which delivers 2mA transcranial direct current stimulation to the primary motor cortex and the dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial direct current stimulation (Nettle device) 2mA stimulation for 20 minutes per day

INTERVENTIONS:
Device: Transcranial direct current stimulation (Nettle device) 2mA stimulation for 20 minutes per day — The Nettle device, manufactured by Samphire Neuroscience, contains four electrodes, two of which provide stimulation to the primary motor cortex (M1), and two stimulate the dorsolateral prefrontal cortex (DLPFC). A treatment session consists of 2mA stimulation for 20 minutes per day. Nettle is a Class IIa medical device which has a CE mark and is currently marketed for use in dysmenorrhoea and the mood component of premenstrual syndrome.

SUMMARY:
Migraine affects 1 in 7 people worldwide, but for those suffering from chronic migraine there is a need for safe, effective and well tolerated treatments. The Nettle device is a non-invasive device, which is worn like a headband and delivers electrical stimulation (known as transcranial direct current stimulation or TCDS) to areas of the brain known to be involved in the processing of pain. In this study, 20 patients will be trained on how to use the device and then use it daily at home for 20 minutes for three months. Patients will complete a headache diary and quality of life questionnaires before using the device, during and after. As this is a feasibility study, adherence to completing the diaries and questionnaires will be assessed. Compliance with the treatment paradigm will also be assessed.

DETAILED DESCRIPTION:
This study is being performed in patients with chronic migraine (CM) which represents a significant burden to both individuals, but also the healthcare system and wider economy. Pharmacological options for the treatment of migraine have expanded in recent years, however, these are not infrequently associated with side effects and are not always effective for all patients. There is an increased need for non-pharmacological treatments such as neuromodulation. Furthermore, non-invasive neuromodulation is relatively safe and, in the case of the Nettle device, can be used at home after a single training session, potentially reducing the burden on healthcare services and increasing patients' autonomy with regards to their treatment.

Transcranial direct current stimulation (tDCS) is a form of non-invasive neuromodulation for which there is an increasing body of evidence in a number of fields including major psychiatric disorders, Parkinson's disease, post-stroke rehabilitation and epilepsy.12,13 The Nettle device, manufactured by Samphire Neuroscience, contains four electrodes, two of which provide stimulation to the primary motor cortex (M1), and two stimulate the dorsolateral prefrontal cortex (DLPFC). A treatment session consists of 2mA stimulation for 20 minutes per day. Nettle is a Class IIa medical device which has a CE mark and is currently marketed for use in dysmenorrhoea and the mood component of premenstrual syndrome. The proposed study would be the first to use Nettle in chronic migraine, therefore a small feasibility study is planned.

The research question is as follows: Is a randomised controlled trial of 12 weeks concurrent M1 and DLPFC tDCS (using the Nettle device) feasible in patients with chronic migraine, with specific regard to recruitment, adherence and monitoring?

The primary objective is: To assess the feasibility of home-based self-administration of tDCS for the preventative treatment of chronic migraine by evaluating recruitment rate, treatment adherence and diary data completeness

The secondary objectives are:

* To generate preliminary estimates of clinical effect size
* To assess tolerability and usability of the Nettle device
* To characterise the safety profile of the Nettle device

The progression criteria are as follows:

* Green (all primary feasibility endpoints met): proceed to definitive randomised controlled trial (RCT) if:

  * Recruitment rate >1 participants per site per month AND
  * Adherence rate ≥75% of schedule tDCS sessions completed AND
  * Diary data completeness >80% of treatment phase days recorded.
* Amber (exactly one primary feasibility endpoint partially met, as defined below): review and refine study processes (e.g. recruitment material, device training, follow up procedures, data-capture methods) and consider repeating feasibility assessment if necessary before proceeding to RCT, if:

  * Recruitment rate 0.8-1.0 participants per site per month
  * Adherence rate 60-75% of scheduled tDCS sessions completed
  * Diary data completeness 65-80% of treatment phase days recorded
* Red (two or more primary feasibility end points unmet, as defined below): halt progression and undertake significant protocol redesign before further feasibility testing

  * Recruitment rate <0.8 participants per site per month
  * Adherence rate <60% of scheduled tDCS sessions completed
  * Diary data completeness <65% of treatment phase days recorded

This is an open label, single arm feasibility study which will be carried out at a single centre. The patients will be primarily recruited from the headache clinic at UCL Queen Square Institute of Neurology. This is expected to generate an ample number of suitable candidates, however additional patients may be recruited from the private headache clinic or via advertisements in migraine charities or support groups.

Appointment one is a virtual appointment to carry out screening (including collecting baseline data as detailed in 7.3.1), electronic written informed consent, carry out quality of life, anxiety and depression questionnaires and to give the patient the headache diary/assist with downloading the Headache Pro App to complete for the following month. If patients are unable to carry out this appointment virtually, they can be offered a face-to-face visit. The virtual or face to face appointment will be carried out by the sub-investigator.

Appointment two is a face-to-face appointment, at least four weeks after the screening appointment at the Queen Square Private Consulting Rooms with the sub-investigator. This visit marks the start of the treatment phase. The following activities are carried out:

* Review of written informed consent and eligibility criteria
* Review of Headache Pro App or paper diary
* Downloading of Nettle App (a representative from Samphire may attend to help troubleshoot)
* Demonstration of the device and explanation of its daily use
* Arrange time and date for final follow up Appointment three is a telephone call from the sub-investigator, one week into the treatment phase, to ensure participants are able to use the device correctly and are completing the diary. For participants using the Headache Pro App, data can be reviewed remotely by the chief investigator. Adverse events are recorded.

Appointment four is a face to face, or virtual visit, three months after the commencement of the treatment phase. The sub-investigator will repeat the quality of life and anxiety and depression questionnaires, ensure headache diaries are completed and review for any adverse events. Adherence will be reviewed (completed sessions are visible on the Samphire App). The patient satisfaction survey is completed at this visit.

Participants are encouraged to contact the sub-investigator between visits, should they develop adverse events, device malfunction, new medication problems which may affect eligibility or any other concern.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 years
2. Fulfil the International Classification of Headache Disorders -3 (ICHD-3) criteria for chronic migraine, diagnosed by a headache specialist, at least 1 year prior to entering the trial
3. Subject is willing to keep headache medications stable for two weeks prior to entering the study and for the duration of the study.
4. Access to a smart phone to use the mobile application to control the device and use the Headache Pro app to record headaches. A paper diary may be used instead of the Headache Pro app Id required by individual patients.
5. Subject is able to provide written informed consent prior to participation in the study
6. Females of childbearing potential agree to use an effective method of contraception from the time consent is signed until treatment discontinuation. Effective methods of contraception acceptable for this trial are the oral contraceptive pill, patch, implant, injection, ring, intra-uterine system, copper coil, barrier methods, partner vasectomy or abstinence. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
7. If there is any possibility of pregnancy, females of childbearing potential should have a negative pregnancy test within 7 days of commencing the treatment phase.
8. Subject must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Epilepsy or history of seizures
2. Current or planned pregnancy during the study timeframe
3. Active suicidal thoughts
4. Pre-existing neurological or neuropsychiatric condition
5. Lesion, tumour or other defect in skull or brain
6. Implant inside skill, cochlear implant or implanted hearing aid.
7. Implanted medical device e.g. pacemaker or neurostimulator
8. Use of other stimulation devices such as spinal cord stimulators, vagal nerve stimulation, auricular nerve stimulator or deep brain stimulation.
9. Concurrent medication overuse
10. Use of cranial botulinum toxin injections or CGRP inhibitors in the past 6 months
11. Current or recent (within three months) participation in another clinical trial.
12. Planned surgical or significant medical intervention during the study period which may affect the study results, at the discretion of the chief investigator.
13. Lacking mental capacity to give informed written consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Average number of participants enrolled per site per month
Adherence rate | 12 weeks
  defined as the proportion of schedule transcranial direct current stimulation sessions completed by each participant
Data completeness | 12 weeks
  defined as the proportion of days with a completed headache diary entry during the 12 week treatment phase

SECONDARY OUTCOMES:
30% responder rate | 12 weeks
  The proportion of patients achieving ≥30% reduction in monthly migraine days (30% responder rate)
Moderate to severe headache days | 12 weeks
  Mean change in monthly number of moderate to severe headache days
Headache Intensity | 12 weeks
  Mean change in monthly headache intensity (on a 0-10 visual analogue scale, with 0 being pain free and 10 being the most severe pain)
Adverse effects | 12 weeks
  Proportion of patients reporting device-related adverse events, with severity grading
Tolerability and usability | 12 weeks
  Patient reported tolerability and usability of the Nettle device, with each item assessed by a Likert 1-5 scale questionnaire as follows:
  1. strongly disagree
  2. somewhat disagree
  3. neither agree nor disagree
  4. somewhat agree
  5. strongly agree
50% responder rate in monthly migraine days | 12 weeks
  Proportion of patients achieving ≥50% reduction in monthly migraine days
30% responder rate for monthly headache days | 12 weeks
  proportion of patients achieving ≥30% reduction in monthly headache days
50% responder rate for monthly headache days | 12 weeks
  proportion of patients achieving 50% reduction in monthly headache days
Change in hospital anxiety scores | 12 weeks
  Mean change in hospital anxiety scores (HADS-A) compared to baseline. HADS-A is scored on a 0-21 scale with 21 being most severe symptoms.
Change in hospital depression score | 12 weeks
  Mean change in hospital depression scores (HADS-D) compared to baseline. HADS-D is scored on a 0-21 scale, with 21 being the most severe symptoms.
Change in migraine disability assessment score | 12 WEEKS
  Mean change in migraine disability assessment score (MIDAS). MIDAS is scored on a 0-270 scale, with higher scores corresponding to more severe symptoms.
Change in headache impact test 6 score (HIT-6) | 12 weeks
  Mean change in HIT6 score compared to baseline. HIT-6 is scored on a 36-78 scale, with higher scores indicating more severe symptoms.
Change in quality of life score | 12 weeks
  Mean change in EuroQol (EQ-5D-5L) quality of life score compared to baseline

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available at reasonable request
Access Criteria: Beginning 12 months after the end point of the trial and ending 3 years after the publication of results.